CLINICAL TRIAL: NCT00483548
Title: A Six-Week, Double-Blind, Multicenter, Placebo Controlled Study Evaluating The Efficacy And Safety Of Flexible Doses Of Oral Ziprasidone As Add-On, Adjunctive Therapy With Lithium, Valproate Or Lamotrigine In Bipolar I Depression
Brief Title: Adjunctive Ziprasidone in the Treatment of Bipolar I Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1281158
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder; Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ziprasidone (Experimental): Active treatment, double-blind, randomized treatment arm
  Interventions: Drug: Ziprasidone
- Placebo (Placebo Comparator): Inactive, placebo treatment, double-blind, randomized arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ziprasidone — Oral capsule formulation to be administered every day for duration of patient's participation in the trial - 40 mg on Day 1; 40 mg twice a day (BID) on Day 2; Flexible BID dosing of 40 mg, 60 mg, 80 mg, 100 mg, 120 mg, 140 mg or 160 mg total daily dose from Day 3 through Week 6. Dose increases of up to 40 mg/day can occur after subject has received previous lower dose for at least 1 day.
  Other Names: Geodon, Zeldox
  Arms: Ziprasidone
Drug: Placebo — Matching placebo oral capsules to be administered as per the instructions for the ziprasidone arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a treatment regimen of ziprasidone plus a mood stabilizer is safe and effective in the short term treatment of Bipolar I Depression. Ziprasidone will be added to lithium, valproate or lamotrigine after the patient has been on a therapeutic dose of one of these mood stabilizers for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for Bipolar I disorder, most recent episode depressed, with or without rapid cycling and without psychotic features. Subjects receive therapeutic dose of lithium, valproate or lamotrigine for at least 4 weeks prior to randomization.

Exclusion Criteria:

* Patients with ultra-fast rapid cycling (8 or more mood episodes per year)
* Significant heart disease including abnormalities in the heart's rhythm (QT prolongation)
* Psychotic symptoms (hallucinations and/or delusions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (53):
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Springdale, Arkansas
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Sanford, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Watertown, Massachusetts
  - Pfizer Investigational Site, Clinton Township, Michigan
  - Pfizer Investigational Site, Saint Charles, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Cherry Hill, New Jersey
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Glen Oaks, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Olean, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Richland, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Brown Deer, Wisconsin
- Australia (4):
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Everton Park, Queensland
  - Pfizer Investigational Site, Spring Hill, Queensland
  - Pfizer Investigational Site, Richmond, Victoria
- India (5):
  - Pfizer Investigational Site, Ellisbridge, Ahmedabad
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Aurangabad, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Delhi, New Delhi

REFERENCES:
- [Derived] Sachs GS, Ice KS, Chappell PB, Schwartz JH, Gurtovaya O, Vanderburg DG, Kasuba B. Efficacy and safety of adjunctive oral ziprasidone for acute treatment of depression in patients with bipolar I disorder: a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Oct;72(10):1413-22. doi: 10.4088/JCP.09m05934. PMID 21672493
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281158&StudyName=Adjunctive%20Ziprasidone%20in%20the%20Treatment%20of%20Bipolar%20I%20Depression

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone; Placebo: Day 1: single dose of 40 milligrams (mg) by mouth (PO); Day 2: 40 mg po twice a day (BID); Day 3 through Week 6: flexible BID dosing titrated to a total daily dose of 40 mg, 60 mg, 80 mg, 100 mg, 120 mg, 140 mg, or 160 mg as adjunctive therapy with a mood stabilizer (lithium, valproate, or lamotrigine).
Period: Overall Study
Arm/Group | Ziprasidone | Placebo
Started | 148 | 150
Received Study Treatment | 147 (1 subject randomized but lost to follow up; no treatment data.) | 147 (3 subjects randomized but not treated.)
Completed | 88 | 104
Not Completed | 60 | 46
Not completed — Randomized; not treated with study drug | 1 | 3
Not completed — Adverse Event | 25 | 14
Not completed — Laboratory abnormality | 1 | 2
Not completed — Lack of Efficacy | 4 | 8
Not completed — Protocol Violation | 11 | 7
Not completed — Pregnancy | 1 | 0
Not completed — Protocol required discontinuation | 6 | 6
Not completed — Unable to comply with protocol schedule | 1 | 0
Not completed — Non-compliance with medication | 2 | 0
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone | Placebo | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 147 | 146 | 293
  >65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 91 | 180
  Male | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts); rated on a 7-point Likert scale 0 (normal) to 6 (most abnormal); total score 0 to 44 (higher score indicates greater severity of symptoms). Change calculated as a difference between post-baseline observation and baseline MADRS score values.
Time Frame: Baseline, Week 6
Population: Intent to Treat analysis set (ITT): all randomized subjects who received at least 1 dose of double-blind treatment and had at least 1 post-baseline primary efficacy evaluation.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale | -14.7 (10.7) | -13.2 (10.4)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; N=141 per arm (282 total) needed for 85% power for 2-sided alpha=0.05 based on true mean difference=4.0 and standard deviation (SD)=11.0 for primary endpoint. Interim Analysis (IA) planned when 60% of subjects had completed study or discontinued prematurely to assess efficacy (nominal 2-sided p-value less than or equal to [≤] 0.0076) or futility (nominal 2-sided p-value greater than or equal to [≥] 0.5099); Test type: Superiority or Other; p = 0.7921, ANCOVA Mixed-effects repeated-measures — Due to planned interim analysis of primary endpoint, to control type I error at 2-sided alpha=0.05, a nominal 2-sided p-value ≤0.0476 needed at final analysis to reject the null hypothesis of no treatment effect; No other adjustment made for multiple comparisons since all comparisons, except for single primary comparison, are considered secondary; Least squares mean = -0.36, 95% CI [-3.07 to 2.34], Standard Error of Mean 1.37 — Mixed-effects repeated-measures (MMRM) analysis of covariance model: fixed categorical effects of treatment, country, mood stabilizer type, visit, treatment-by-visit interaction, fixed continuous effect of baseline value and subject as random effect

2. Secondary Outcome: Change From Baseline to Week 6 in Clinical Global Impression - Severity Scale (CGI-Severity or CGI-S)
Description: CGI-S is a single-item clinician rated scale used to assess global severity of bipolar illness based on an overall evaluation of symptoms of bipolar mania, associated behavioral symptoms, and condition of the subject. Scored from 1 (normal, not at all ill) to 7 (among the most severely ill subjects). Higher score = more affected. Change calculated as a difference between post-baseline observation and baseline CGI-S score values.
Time Frame: Baseline, Week 6
Population: ITT
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale | -1.5 (1.3) | -1.5 (1.2)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 6; MMRM analysis of covariance model with fixed categorical effects of treatment, country, type of mood stabilizer, visit, treatment-by-visit interaction, fixed continuous effect of baseline value and subject as random effect; Test type: Superiority or Other; p = 0.7223, ANCOVA Mixed-effects repeated-measures; Least squares mean = 0.06, 95% CI [-0.25 to 0.36], Standard Error of Mean 0.16

3. Secondary Outcome: MADRS Remission: Number of Subjects With Total MADRS Score ≤ 12 at Week 6
Description: Number of subjects with MADRS total score ≤ 12 (indicates remission). MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts); rated on a 7-point Likert scale 0 (normal) to 6 (most abnormal); total score 0 to 44 (higher score indicates greater severity of symptoms).
Time Frame: Week 6
Population: ITT; Last observation carried forward (LOCF)
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
participants | 48 | 54
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 6; LOCF; Logistic regression model with treatment, country, and type of mood stabilizer; Test type: Superiority or Other; p = 0.5029, Regression, Logistic; Odds Ratio (OR) = 0.846, 95% CI [0.52 to 1.38] — Odds ratio measures the odds of achieving remission (MADRS total score ≤ 12) from ziprasidone treated subjects versus placebo; a value > 1 favors ziprasidone

4. Secondary Outcome: MADRS Response: Number of Subjects With Total MADRS Score Reduction ≥ 50 Percent From Baseline at Week 6
Description: Number of subjects with reduction of ≥50 percent (%) in MADRS total score (indicates response). MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts); rated on a 7-point Likert scale 0 (normal) to 6 (most abnormal); total score 0 to 44 (higher score indicates greater severity of symptoms). Reduction calculated as ([A-B]/B*100): A=value at observation; B=baseline value.
Time Frame: Week 6
Population: ITT; LOCF
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
participants | 62 | 65
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 6; LOCF; Logistic regression model with treatment, country, and type of mood stabilizer; Test type: Superiority or Other; p = 0.8266, Regression, Logistic; Odds Ratio (OR) = 0.949, 95% CI [0.59 to 1.52] — Odds ratio measures the odds of achieving response (≥ 50 % reduction in MADRS total score) from ziprasidone treated subjects versus placebo; a value > 1 favors ziprasidone

5. Secondary Outcome: Clinical Global Impression - Improvement Scale (CGI-Improvement or CGI-I): Number of Subjects With Response (Much Improved or Very Much Improved) at Week 6
Description: Number of subjects with improvement defined as CGI-I response of 1 (very much improved) or 2 (much improved). CGI-I is a single-item clinician rated scale used to assess global improvement in the subject's clinical state (bipolar mania) in response to study treatment and as compared to their status at pre-treatment baseline. Scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse). Higher score = more affected.
Time Frame: Baseline, Week 6
Population: ITT; LOCF
Measure: Number; unit: participants
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
participants | 66 | 69
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 6; LOCF; Logistic regression model with treatment, country, and type of mood stabilizer; Test type: Superiority or Other; p = 0.7924, Regression, Logistic — Logistic regression model with treatment, country, and type of mood stabilizer; Odds Ratio (OR) = 0.939, 95% CI [0.59 to 1.50]

6. Secondary Outcome: Change From Baseline in MADRS Total Score (Post-baseline Excluding Week 6)
Description: as for outcome 1
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5
Population: ITT; LOCF; (n)=number of subjects with analyzable data: baseline and post-baseline observation for ziprasidone, placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 1 (n=142, 141) | -8.1 (7.9) | -6.1 (7.3)
  Week 2 (n=121, 139) | -11.7 (8.9) | -9.0 (8.6)
  Week 3 (n=115, 130) | -13.0 (9.5) | -11.0 (9.2)
  Week 4 (n=106, 122) | -14.1 (9.6) | -11.8 (9.5)
  Week 5 (n=103, 112) | -14.9 (9.4) | -13.3 (10.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 1; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0594, ANCOVA; Least squares mean = -1.68, 95% CI [-3.42 to 0.07], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Week 2; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.2230, ANCOVA; Least squares mean = -1.25, 95% CI [-3.27 to 0.77], Standard Error of Mean 1.03
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Week 3; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.6971, ANCOVA; Least squares mean = -0.43, 95% CI [-2.57 to 1.72], Standard Error of Mean 1.09
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Week 4; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.5485, ANCOVA; Least squares mean = -0.68, 95% CI [-2.89 to 1.54], Standard Error of Mean 1.12
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; Week 5; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.8322, ANCOVA; Least squares mean = -0.25, 95% CI [-2.60 to 2.10], Standard Error of Mean 1.19

7. Secondary Outcome: Change From Baseline in CGI-Severity Score (Post-baseline Excluding Week 6)
Description: CGI-S is a single-item clinician rated scale used to assess global severity of bipolar illness based on an overall evaluation of symptoms of bipolar mania, associated behavioral symptoms, and condition of the subject. Scores range from 1 (normal, not at all ill) to 7 (among the most severely ill subjects). Higher score = more affected. Change calculated as a difference between post-baseline observation and baseline CGI-S score values.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 1 (n=142, 141) | -0.5 (0.8) | -0.4 (0.8)
  Week 2 (n=120, 139) | -0.9 (1.1) | -0.7 (0.9)
  Week 3 (n=115, 130) | -0.9 (1.0) | -0.9 (1.0)
  Week 4 (n=106, 122) | -1.1 (1.1) | -1.1 (1.1)
  Week 5 (n=103, 112) | -1.3 (1.2) | -1.3 (1.2)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1771, ANCOVA; Least squares mean = -0.12, 95% CI [-0.29 to 0.05], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.1765, ANCOVA; Least squares mean = -0.15, 95% CI [-0.37 to 0.07], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.6765, ANCOVA; Least squares mean = -0.05, 95% CI [-0.27 to 0.18], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.9770, ANCOVA; Least squares mean = 0.00, 95% CI [-0.24 to 0.25], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.7907, ANCOVA; Least squares mean = -0.04, 95% CI [-0.30 to 0.23], Standard Error of Mean 0.13

8. Secondary Outcome: CGI-Improvement Score
Description: CGI-I is a single-item clinician rated scale used to assess global improvement in the subject's clinical state (bipolar mania) in response to study treatment and as compared to their status at pre-treatment baseline. Scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse). Higher score = more affected. Week 6 is the primary timepoint.
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: ITT; LOCF; (n)=number of subjects with analyzable data at baseline and post-baseline observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 1 (n=142, 141) | 3.2 (0.9) | 3.4 (0.8)
  Week 2 (n=120, 138) | 2.9 (1.1) | 3.1 (1.0)
  Week 3 (n=115, 130) | 2.7 (1.0) | 2.9 (1.0)
  Week 4 (n=106, 122) | 2.6 (1.2) | 2.8 (1.2)
  Week 5 (n=103, 112) | 2.5 (1.2) | 2.6 (1.1)
  Week 6 (n=92, 108) | 2.4 (1.2) | 2.4 (1.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 1; LOCF; Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Test type: Superiority or Other; p = 0.0392, ANOVA; Least squares mean = -0.22, 95% CI [-0.43 to -0.01], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Week 2; LOCF; Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Test type: Superiority or Other; p = 0.2803, ANOVA; Least squares mean = -0.14, 95% CI [-0.38 to 0.11], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Week 3; LOCF; Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Test type: Superiority or Other; p = 0.9835, ANOVA; Least squares mean = -0.00, 95% CI [-0.26 to 0.26], Standard Error of Mean 0.13
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Week 4; LOCF; Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Test type: Superiority or Other; p = 0.7062, ANOVA; Least squares mean = -0.06, 95% CI [-0.34 to 0.23], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; Week 5; LOCF; Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Test type: Superiority or Other; p = 0.9518, ANOVA; Least squares mean = -0.01, 95% CI [-0.31 to 0.29], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; Week 6; LOCF; Test type: Superiority or Other; p = 0.4757, ANOVA — Analysis of variance model with treatment, country, type of mood stabilizer as fixed effects; Least squares mean = 0.11, 95% CI [-0.20 to 0.42], Standard Error of Mean 0.16

9. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score
Description: HAM-A is a clinician rated 14-item scale that rates the intensity of psychic anxiety (items 1 to 6 and item 14) and somatic anxiety (items 7 to 13) on a 5-point severity scale; scores range from 0 (not present) to 4 (very severe); lower score indicates less affected. Change calculated as a difference between post-baseline observation and baseline HAM-A score values. Week 6 is the primary timepoint.
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 2 (n=136, 141) | -5.6 (6.8) | -5.9 (6.7)
  Week 4 (n=111, 127) | -7.1 (7.2) | -7.4 (7.6)
  Week 6 (n=100, 111) | -8.5 (7.9) | -8.6 (7.5)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.6362, ANCOVA; Least squares mean = 0.35, 95% CI [-1.12 to 1.82], Standard Error of Mean 0.75
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.4565, ANCOVA; Least squares mean = 0.59, 95% CI [-0.98 to 2.17], Standard Error of Mean 0.80
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Week 6; LOCF; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.4770, ANCOVA; Least squares mean = 0.61, 95% CI [-1.08 to 2.30], Standard Error of Mean 0.86

10. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score
Description: YMRS is clinician rated 11-item scale (elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, speech [rate and amount], language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight) used to assess the severity of manic symptoms and effect of treatment on mania severity. Seven items ranked on scale from 0 to 4; 4 items ranked 0 to 8. Higher scores indicate greater severity. Change calculated as a difference between post-baseline observation and baseline YMRS score values. Week 6 is the primary timepoint.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 1 (n=142, 141) | 0.7 (4.4) | -0.2 (3.5)
  Week 2 (n=121, 139) | 0.5 (4.5) | -0.2 (4.3)
  Week 3 (n=115, 130) | -0.0 (4.5) | -0.2 (4.9)
  Week 4 (n=106, 122) | -0.9 (4.1) | -1.1 (4.2)
  Week 5 (n=103, 112) | -0.9 (3.9) | -1.3 (4.1)
  Week 6 (n=92, 108) | -1.0 (4.8) | -0.9 (4.6)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1277, ANCOVA; Least squares mean = 0.70, 95% CI [-0.20 to 1.60], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p = 0.2345, ANCOVA; Least squares mean = 0.64, 95% CI [-0.41 to 1.68], Standard Error of Mean 0.53
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.8337, ANCOVA; Least squares mean = 0.13, 95% CI [-1.05 to 1.30], Standard Error of Mean 0.60
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 4]; Test type: Superiority or Other; p = 0.4646, ANCOVA; Least squares mean = 0.43, 95% CI [-0.73 to 1.59], Standard Error of Mean 0.59
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.3993, ANCOVA; Least squares mean = 0.50, 95% CI [-0.67 to 1.67], Standard Error of Mean 0.59
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 9, analysis 3]; Test type: Superiority or Other; p = 0.7647, ANCOVA; Least squares mean = 0.19, 95% CI [-1.08 to 1.46], Standard Error of Mean 0.65

11. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Scale at Week 6
Description: GAF is a clinician rated scale to measure the severity of illness-related impairment in psychological, social, and occupational functioning using a 100-point scale (single score of 1 to 100) with 100 indicating a superior level of function. Change calculated as a difference between post-baseline observation and baseline GAF score values.
Time Frame: Baseline, Week 6
Population: ITT; observed cases; Early Termination (ET) visits re-slotted to regular weekly visits according to duration since first dosing date; ET Visit only includes observations from visits that did not meet windowing criteria; (n)=number of subjects with analyzable data at baseline and post-baseline observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 6 (n=100, 110) | 14.7 (13.8) | 11.2 (12.3)
  ET (n=34, 27) | 0.0 (7.1) | 2.8 (9.1)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0108, ANCOVA; Least squares mean = 4.24, 95% CI [0.99 to 7.50], Standard Error of Mean 1.65

12. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Week 6 (Items 1 Through 3)
Description: SDS is a 5-item subject rated scale to measure the extent to which work and or school, social life and or leisure activities, and home life and or family responsibilities were impaired by psychiatric illness. Items 1 to 3 rated on 11-point scale ranging 0 (not at all) to 10 (extremely affected). Total score 0 to 30; higher score indicates greater impairment; items 4 and 5 report number of days in the last month (0 to 31) subject missed work or school or was unproductive and are rated separately. Change calculated as a difference between post-baseline observation and baseline SDS score values.
Time Frame: Baseline, Week 6
Population: ITT; ET visits re-slotted to regular weekly visits according to duration since first dosing date; ET Visit only includes observations from visits that did not meet windowing criteria; (n)=number of subjects with analyzable data at baseline and post-baseline observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Total SDS: Week 6 (n=58, 63) | -8.5 (9.2) | -3.7 (8.2)
  Total SDS: ET (n=19, 14) | 0.2 (6.8) | -1.4 (6.7)
  Work/School: Week 6 (n=58, 64) | -2.1 (3.5) | -1.6 (2.9)
  Work/School: ET (n=19, 14) | 0.4 (3.0) | -0.1 (2.7)
  Social life: Week 6 (n=94, 102) | -2.5 (3.3) | -1.7 (3.2)
  Social life: ET (n=31, 23) | -0.5 (2.9) | 0.1 (3.1)
  Family/Home: Week 6 (n=94, 102) | -2.6 (3.2) | -1.7 (3.3)
  Family/Home: ET (n=31, 23) | 0.2 (2.3) | -0.6 (3.2)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Total SDS: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0010, ANCOVA; Least squares mean = -4.56, 95% CI [-7.24 to -1.87], Standard Error of Mean 1.35

13. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Week 6 (Items 4 and 5)
Description: as for outcome 12
Time Frame: Baseline, Week 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
days
  Days lost: Week 6 (n=85, 93) | -1.2 (2.5) | -0.7 (2.3)
  Days lost: ET (n=29, 21) | 0.5 (2.7) | 0.0 (2.2)
  Days unproductive: Week 6 (n=87, 89) | -1.6 (2.8) | -1.3 (2.9)
  Days unproductive: ET (n=29, 21) | -0.2 (2.5) | -0.1 (3.7)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Days Lost: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.1230, ANCOVA; Least squares mean = -0.44, 95% CI 2-sided [-1.00 to 0.12], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Days Unproductive: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.6232, ANCOVA; Least squares mean = -0.17, 95% CI 2-sided [-0.84 to 0.50], Standard Error of Mean 0.34

14. Other Pre Specified Outcome: Change From Baseline in Simpson Angus Scale (SAS) Score
Description: SAS is a clinician rated 10-item scale to measure extrapyramidal side effects (Parkinsonism or Parkinsonian side effects induced with antipsychotics); rated on a 5-point scale with range 0 (absence of condition) to 4 (presence of condition in extreme form). Global score is sum of all scores divided by the total number of items. Change calculated as a difference between post-baseline observation and baseline SAS score values.
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: ITT; (n)=number of subjects with analyzable data at baseline and post-baseline observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 2 (n=136, 141) | 0.1 (0.8) | -0.1 (0.7)
  Week 4 (n=111, 126) | 0.0 (0.8) | 0.0 (0.6)
  Week 6 (n=100, 110) | 0.0 (0.7) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Week 2; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0096, ANCOVA; Least squares mean = 0.17, 95% CI [0.04 to 0.31], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Week 4; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.8134, ANCOVA; Least squares mean = 0.02, 95% CI [-0.13 to 0.16], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.0226, ANCOVA; Least squares mean = 0.16, 95% CI [0.02 to 0.29], Standard Error of Mean 0.07

15. Other Pre Specified Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS or BAS)
Description: BARS is a clinician rated scale to evaluate akathisia associated with use of antipsychotic medications: objective motor restlessness, range 0 to 3; subjective complaints of restlessness and associated distress, range 0 to 3; global clinical assessment of akathisia, range 0 to 5. Higher scores indicate more affected. Change calculated as a difference between post-baseline observation and baseline BARS score values.
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: ITT; Summarized as Global BARS; individual scores not summarized; (n)=number of subjects with analyzable data at observation for ziprasidone and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Week 2 (n=135, 139) | 0.1 (0.5) | -0.0 (0.4)
  Week 4 (n=111, 125) | 0.0 (0.5) | 0.0 (0.5)
  Week 6 (n=100, 110) | 0.0 (0.6) | -0.0 (0.5)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0193, ANCOVA; Least squares mean = 0.12, 95% CI [0.02 to 0.23], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.4745, ANCOVA; Least squares mean = 0.04, 0.16% CI [-0.07 to 0.16], Standard Error of Mean 0.06
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2613, ANCOVA; Least squares mean = 0.07, 95% CI [-0.05 to 0.19], Standard Error of Mean 0.06

16. Other Pre Specified Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Scores
Description: AIMS is a clinician rated 12-item scale to rate 7 body areas and global judgments on the severity of abnormal movements, incapacitation and subject's awareness of abnormal movements. Items 1 to 10 scored 0 (none) to 4 (severe); items 11 to 14 are No or Yes response to dental status and sleep movements and are assessed separately. AIMS total score is sum of first 7 items. Change calculated as a difference between post-baseline observation and baseline AIMS score values.
Time Frame: Baseline, Week 2, Week 4, Week 6
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Total score: Week 2 (n=136, 142) | 0.1 (0.7) | -0.1 (0.4)
  Total score: Week 4 (n=111, 127) | -0.0 (0.5) | -0.0 (0.5)
  Total score: Week 6 (n=100, 111) | -0.0 (0.6) | -0.0 (0.4)
  Global severity score: Week 2 (n=136, 142) | 0.0 (0.4) | -0.0 (0.2)
  Global severity score: Week 4 (n=111, 127) | 0.0 (0.3) | 0.0 (0.2)
  Global severity score: Week 6 (n=100, 111) | 0.0 (0.3) | 0.0 (0.1)
  Incapacitation score: Week 2 (n=136, 142) | 0.0 (0.2) | -0.0 (0.1)
  Incapacitation score: Week 4 (n=111, 127) | 0.0 (0.1) | -0.0 (0.2)
  Incapacitation score: Week 6 (n=100, 111) | 0.0 (0.1) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Total score: Week 2; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0271, ANCOVA; Least squares mean = 0.11, 95% CI [0.01 to 0.21], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Total score: Week 4; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.7462, ANCOVA; Least squares mean = -0.01, 95% CI [-0.07 to 0.05], Standard Error of Mean 0.03
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Total score: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.9574, ANCOVA; Least squares mean = 0.00, 95% CI [-0.08 to 0.08], Standard Error of Mean 0.04
Statistical Analysis 4: Comparison: Ziprasidone vs Placebo; Global severity score: Week 2; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.0844, ANCOVA; Least squares mean = 0.05, 95% CI [-0.01 to 0.10], Standard Error of Mean 0.03
Statistical Analysis 5: Comparison: Ziprasidone vs Placebo; Global severity score: Week 4; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.5779, ANCOVA; Least squares mean = 0.01, 95% CI [-0.04 to 0.06], Standard Error of Mean 0.02
Statistical Analysis 6: Comparison: Ziprasidone vs Placebo; Global severity score: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.7455, ANCOVA; Least squares mean = 0.01, 95% CI [-0.05 to 0.06], Standard Error of Mean 0.03
Statistical Analysis 7: Comparison: Ziprasidone vs Placebo; Incapacitation score: Week 2; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.3278, ANCOVA; Least squares mean = 0.02, 95% CI [-0.02 to 0.05], Standard Error of Mean 0.02
Statistical Analysis 8: Comparison: Ziprasidone vs Placebo; Incapacitation score: Week 4; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.9097, ANCOVA; Least squares mean = 0.00, 95% CI [-0.03 to 0.03], Standard Error of Mean 0.01
Statistical Analysis 9: Comparison: Ziprasidone vs Placebo; Incapacitation score: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.9864, ANCOVA; Least squares mean = 0.00, 95% CI [-0.04 to 0.04], Standard Error of Mean 0.02

17. Secondary Outcome: Change From Baseline in Quality of Life, Enjoyment, and Satisfaction Scale (Q-LES-Q) Scores at Week 6
Description: Q-LES-Q is a 16-item subject rated scale to measure satisfaction with areas of daily functioning (physical health, social relationships, medication, and overall life satisfaction); rated on a 5-point Likert scale: higher scores indicate greater enjoyment and satisfaction with general life activities. Scores for items 1 to 14 are summed for a total score and converted to 0 to 100 range. Items 15 and 16 measure satisfaction with medication and overall satisfaction and are analyzed separately. Change calculated as a difference between post-baseline observation and baseline Q-LES-Q score values.
Time Frame: Baseline, Week 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Ziprasidone | Placebo
Number analyzed (Participants) | 145 | 145
scores on scale
  Total Q-LES-Q: Week 6 (n=82, 94) | 15.2 (19.0) | 11.6 (17.3)
  Total Q-LES-Q: ET (n=27, 17) | -0.1 (19.7) | 1.6 (14.5)
  Medications: Week 6 (n=91, 93) | 0.4 (1.2) | 0.3 (1.1)
  Medications: ET (n=27, 20) | -0.3 (1.2) | -0.4 (0.8)
  Overall life satisfaction: Week 6 (n=94, 103) | 0.8 (1.1) | 0.5 (1.1)
  Overall life satisfaction: ET (n=31, 23) | 0.1 (1.3) | 0.0 (0.9)
Statistical Analysis 1: Comparison: Ziprasidone vs Placebo; Total Q-LES-Q: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.5519, ANCOVA; Least squares mean = 1.52, 95% CI [-3.50 to 6.53], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: Ziprasidone vs Placebo; Medications: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.5238, ANCOVA; Least squares mean = -0.09, 95% CI [-0.35 to 0.18], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Ziprasidone vs Placebo; Overall life satisfaction: Week 6; Observed cases; Analysis of covariance model with treatment, country, type of mood stabilizer as fixed effects and baseline score as covariate; Test type: Superiority or Other; p = 0.5360, ANCOVA; Least squares mean = 0.09, 95% CI [-0.19 to 0.36], Standard Error of Mean 0.14

ADVERSE EVENTS:
Arm/Group | Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 1/147 | 6/147
Other Adverse Events (participants affected / at risk) | 96/147 | 57/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=147) | Placebo (N=147)
Palpitations (Cardiac disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=147) | Placebo (N=147)
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Nausea (Gastrointestinal disorders) | 16 | 8
Fatigue (General disorders) | 19 | 6
Akathisia (Nervous system disorders) | 8 | 2
Dizziness (Nervous system disorders) | 19 | 9
Headache (Nervous system disorders) | 17 | 14
Sedation (Nervous system disorders) | 21 | 7
Somnolence (Nervous system disorders) | 33 | 7
Tremor (Nervous system disorders) | 13 | 10
Anxiety (Psychiatric disorders) | 9 | 1
Insomnia (Psychiatric disorders) | 17 | 10
Restlessness (Psychiatric disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.